CLINICAL TRIAL: NCT00003517
Title: Phase II Study of Antineoplastons A10 and AS2-1 Capsules With Total Androgen Blockade in Patients With Stage III or IV Adenocarcinoma of the Prostate
Brief Title: Antineoplaston Therapy in Treating Patients With Stage III or Stage IV Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-PR-6; CDR0000066560 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Adenocarcinoma of the Prostate; Stage III Prostate Cancer; Stage IV Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1; bicalutamide; Flutamide; Leuprolide; Androgen Antagonists; Biological Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: antineoplaston AS2-1
Drug: bicalutamide
Drug: flutamide
Drug: leuprolide acetate
Procedure: alternative product therapy
Procedure: antiandrogen therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: complementary and alternative therapy
Procedure: differentiation therapy
Procedure: endocrine therapy
Procedure: hormone therapy

SUMMARY:
RATIONALE: Antineoplastons are naturally occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial is studying how well antineoplaston therapy works in treating patients with stage III or stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of antineoplastons A10 and AS2-1 capsules in combination with total androgen blockade in patients with localized, regional or metastatic adenocarcinoma of the prostate by determining the proportion of patients who experience an objective tumor response.
* Evaluate the adverse effects of and tolerance to this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive gradually escalating doses of antineoplastons A10 and AS2-1 capsules orally 6-7 times daily until the maximum tolerated dose is reached. Treatment continues for at least 3 months in the absence of disease progression or unacceptable toxicity. Concurrently, patients continue hormonal therapy with flutamide, leuprolide, or bicalutamide at the same dose as before beginning antineoplaston therapy.

Tumors are measured every 4 months for 2 years, every 6 months for 2 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven localized, regional, or metastatic adenocarcinoma of the prostate
* Progressive disease during prior hormonal therapy (both antiandrogen and gonadotropin-releasing hormone) and must continue hormonal therapy
* Measurable tumors or tumor markers
* Bone metastases allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* No hepatic failure
* Bilirubin no greater than 2.5 mg/dL
* SGOT no greater than 2 times normal

Renal:

* No chronic renal failure
* BUN less than 60 mg/dL
* Creatinine no greater than 2.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* Blood ammonia normal

Cardiovascular:

* No severe heart disease

Pulmonary:

* No severe lung disease

Other:

* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other prior or concurrent second malignancy within the past 2 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* At least 4 weeks since prior investigational clinical trial
* No other concurrent treatment for metastatic prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States